CLINICAL TRIAL: NCT01748266
Title: Interest of the Measure of the StO2 to Estimate the Microcirculatory Disturbances Following Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: Microcirculation of the Thenar Eminence
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1008018; 2010-A00172-37 (Other: ANSM)
Record Dates: First submitted 2012-12-07; First posted 2012-12-12 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Elective Cardiac Surgery
Keywords: StO2; microcirculation; NIRS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- microcirculatory reactivity: Patients were studied during the first 48 postoperative hours. Microcirculation of the thenar eminence was analyzed by NIRS technology, through the StO2 and the resaturation slope after an ischemic challenge.
  Interventions: Other: microcirculatory reactivity

INTERVENTIONS:
Other: microcirculatory reactivity — Microcirculation of the thenar eminence was analyzed by NIRS technology, through the StO2 and the resaturation slope after an ischemic challenge.

SUMMARY:
Microcirculatory disturbances following cardiac surgery with cardiopulmonary bypass (CPB) have been thought to be at the origin of organ dysfunction. Though, few studies correlated microvascular alterations with outcome. Investigators aimed at firstly describing microcirculation with near infra red spectroscopy (NIRS) and secondly correlating NIRS parameters with intensive care length of stay and organ dysfunction.

DETAILED DESCRIPTION:
40 patients at high risk of post operative systemic inflammatory response syndrome after an elective cardiac surgery with CPB were included in this prospective observational study. Patients were studied during the first 48 postoperative hours. Microcirculation of the thenar eminence was analyzed by NIRS technology, through the StO2 and the resaturation slope after an ischemic challenge. Organ dysfunction was assessed with the SOFA score.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* scheduled for an elective cardiac surgery at high risk of post operative systemic inflammatory response syndrome

Exclusion Criteria:

* BMI>35

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients at high risk of post operative systemic inflammatory response syndrome after an elective cardiac surgery with CPB
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
microcirculatory reactivity | 10 minutes before anesthésia induction
  Tissue oxygen saturation (StO2) measure by a tissue spectrometer with a 25 mm probe spacing placed on the thenar eminence

SECONDARY OUTCOMES:
microcirculatory reactivity | during CPB (30 minutes after the start), and 2, 6, 12, 24 and 48 hours after the end of the CPB
  Tissue oxygen saturation (StO2) measure by a tissue spectrometer with a 25 mm probe spacing placed on the thenar eminence

CONTACTS AND LOCATIONS:
Overall Officials: Jerome MOREL, Md, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France